CLINICAL TRIAL: NCT06284902
Title: Open-Label, Single-Dose, Randomized, 6-Treatment, 6-Sequence, 6-Period Crossover Relative Bioavailability Study Comparing Fexofenadine HCl New Formulation Tablets (Test Drug) With or Without Water to Fexofenadine HCl Coated Tablets (Reference Drug) With Water in Healthy Male and Female Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Fexofenadine HCl New Formulation Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opella Healthcare Group SAS, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDR17987
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Treatment Sequence Group 1 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet
- Treatment Sequence Group 2 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet
- Treatment Sequence Group 3 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet
- Treatment Sequence Group 4 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet
- Treatment Sequence Group 5 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet
- Treatment Sequence Group 6 (Experimental)
  Interventions: Drug: Fexofenadine HCl Coated tablet; Drug: Fexofenadine HCl New Formulation Tablet

INTERVENTIONS:
Drug: Fexofenadine HCl Coated tablet — Film-coated tablet.
Drug: Fexofenadine HCl New Formulation Tablet — New formulation tablet.

SUMMARY:
The purpose of the study is to assess the relative bioavailability of a new galenic form of fexofenadine HCl new formulation tablet (test drug) taken with or without water compared to fexofenadine HCl film-coated tablets (reference form) taken with water under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female non-smokers (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤55 years of age, with body-mass-index (BMI) >18 and <29.9 kilogram per meter square (kg/m^2) and body weight ≥50.0 kg to ≤100.0 kg for males and ≥40.0 kg to ≤90.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to inclusion on Day 1.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Standard 12-lead electrocardiogram (ECG) parameters after 5 minutes resting in supine position in the following ranges:120 milliseconds (ms)<PR<220 ms, QRS<120 ms, QTcF≤450 ms if male, ≤470 ms if female and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
4. Female participants of non-childbearing potential must be:

   1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to inclusion on Day 1) with confirmation by documented follicle-stimulating hormone (FSH) levels 30 milli-international units per milliliter (mIU/mL); or
   2. surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy or tubal ligation) at least 3 months prior to inclusion on Day 1.
5. Female participants of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized for at least 3 months prior to inclusion on Day 1) must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last dose:

   1. simultaneous use of hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to inclusion on Day 1 (must agree to use the same contraceptive throughout the study) and condom for the male partner;
   2. simultaneous use of non-hormonal intrauterine device placed at least 4 weeks prior to inclusion on Day 1 and condom for the male partner;
   3. simultaneous use of diaphragm or cervical cap with spermicide and condom for the male partner, started at least 21 days prior to inclusion on Day 1.
6. Male participants who are not vasectomized for at least 3 months prior to inclusion on Day 1 and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from the first dose and for 90 days after the last dose:

   1. simultaneous use of condom and hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;
   2. simultaneous use of condom and a diaphragm or cervical cap with spermicide for the female partner.
7. Male participants (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from the first dose and for 90 days after the last dose.
8. Male participants must be willing not to donate sperm for 90 days after the last dose.
9. Willing to take off dentures or mouth piercing at the time of dosing.
10. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
3. Frequent history of headaches and/or migraine more than twice a month, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
4. Positive pregnancy test or lactating female participant.
5. Positive urine drug screen, urine cotinine test, or alcohol breath test.
6. Known allergic reactions to fexofenadine HCl or other related drugs, or to any excipient in the formulation.
7. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
8. Clinically significant ECG abnormalities or vital signs abnormalities (systolic blood pressure lower than 95 or over 140 mmHg, diastolic blood pressure lower than 45 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
9. Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease of ≥20 mmHg in systolic blood pressure, decrease of ≥10 mmHg in diastolic blood pressure, and increase of ≥30 bpm in heart rate within 3 minutes when changing from supine to standing position.
10. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
11. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
12. Use of medications for the timeframes specified below, with the exception of hormonal contraceptives and medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the pharmacokinetic (PK) profile of the study drug or participant safety (e.g., topical drug products without significant systemic absorption):

    1. any biologics (antibody or its derivatives) given within 4 months prior to inclusion on Day 1;
    2. depot injection or implant within 3 months prior to inclusion on Day 1;
    3. any drug known to induce or inhibit cytochrome P450 (CYP)3A4 metabolism, including St. John's wort, within 30 days prior to inclusion on Day 1;
    4. prescription medications within 14 days prior to inclusion on Day 1;
    5. any vaccine, including COVID-19 vaccine, within 28 days prior to inclusion on Day 1;
    6. over-the-counter (OTC) medications and natural health products (including herbal remedies such as homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to inclusion on Day 1, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    7. any drug known to be P-glycoproteins (Pg-p) inhibitors or inducers, Organic anion transporting polypeptides (OATP) inhibitors or inducers or any medication containing ketoconazole (e.g., Nizoral), itraconazole, verapamil, erythromycin, rifampin, and carbamazepine within 14 days prior to inclusion on Day 1 and during the study period.
    8. any antacids containing aluminum and magnesium within 14 days prior to inclusion on Day 1 and during the study period.
    9. any antihistaminic drug within 14 days prior to inclusion on Day 1.
    10. any tricyclic antidepressants within 14 days prior to inclusion on Day 1.
13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to inclusion on Day 1, administration of a biological product in the context of a clinical research study within 90 days prior to inclusion on Day 1, or concomitant participation in an investigational study involving no drug or device administration.
14. Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
15. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first inclusion on Day 1.
16. Presence of orthodontic braces or orthodontic retention wires or dentures, or any physical findings in the mouth or tongue that would be likely to interfere with successful completion of the dosing procedure.
17. Presents difficulty with venipuncture and/or poor venous access.
18. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero Until the Last Observed Concentration (AUC0-t) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hours (hrs) post-dose
Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) (AUC0-inf) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose
Maximal Observed Concentration (Cmax) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose

SECONDARY OUTCOMES:
Time When the Maximal Concentration is Observed (Tmax) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose
Time of Observation Prior to the First Observation with a Measurable (non-zero) Concentration (Tlag) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose
Terminal Half-life Associated with the Terminal Slope (T1/2z) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose
Terminal Elimination Rate Constant (Kel) of Fexofenadine | Pre-dose and 0.17, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 36.0, and 48.0 hrs post-dose
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | From screening up to 7-10 days post last dose (approximately 13 weeks)
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical trial participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. A TEAE is defined as AEs that occurred or worsened at any time during the on-treatment period are defined as treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Syneos Health Clinic inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BDR17987 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25620&tenant=MT_SNY_9011